CLINICAL TRIAL: NCT06952920
Title: Electroacupuncture for Managing Chemotherapy-Induced Gastrointestinal Symptom Clusters in Patients With Breast Cancer
Brief Title: Electroacupuncture for Chemotherapy-Induced GI Symptom Clusters in Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiuda Zhao (Other)
Responsible Party: Sponsor-Investigator, Jiuda Zhao, Clinical Professor, Affiliated Hospital of Qinghai University
Organization: Affiliated Hospital of Qinghai University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AHQU-2025002
Record Dates: First submitted 2025-04-16; First posted 2025-05-01 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Standard Quadruple Antiemetic Therapy; Electroacupuncture; Chemotherapy-induced Gastrointestinal Symptom Cluster
Keywords: breast cancer; chemotherapy; standard quadruple antiemetic therapy; electroacupuncture; chemotherapy-induced gastrointestinal symptom cluster
MeSH Terms: conditions — Breast Neoplasms | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- true acupuncture + standard quadruple antiemetic therapy (Experimental): The experimental group received electroacupuncture (EA) combined with a standard quadruple antiemetic regimen comprising Olanzapine (2.5 mg orally daily, days 1-4), dexamethasone (10 mg intravenously day 1; 7.5 mg intravenously days 2-3), a 5-HT₃ antagonist (palonosetron 0.25 mg intravenously or 0.5 mg orally, or ondansetron 8 mg intravenously or 8 mg orally twice, or tropisetron 5 mg intravenously, all on day 1), and an NK₁ antagonist (fosaprepitant 150 mg intravenously, or aprepitant 130 mg intravenously, or oral aprepitant 125 mg day 1 then 80 mg days 2-3, or netupitant 300 mg orally day 1). EA was applied at Zusanli (ST36), Neiguan (PC6), Hegu (LI4), and Zhaohai (KI6) with insertion depths of 20 mm, 15 mm, 20 mm, and 5 mm respectively, using continuous wave mode at 2 Hz and current intensity ≤10 mA (tolerance-adjusted) for 30 minutes per session. Treatment started 1-2 hours pre-chemotherapy on day 1 and continued daily at 9:00-10:00 on days 2-4, totaling four sessions per cycle.
  Interventions: Device: electroacupuncture; Drug: standard quadruple antiemetic therapy
- sham acupuncture + standard quadruple antiemetic therapy (Placebo Comparator): The control group received sham electroacupuncture combined with the identical standard quadruple antiemetic regimen (drug components and dosages identical to the experimental group). The sham intervention protocol consisted of: (1) superficial needle insertion at non-acupoint locations adjacent to the authentic acupoints (ST36, PC6, LI4, and KI6); (2) attachment of non-functional electrodes using deactivated electroacupuncture devices with identical appearance to active units; while maintaining identical treatment duration (30 minutes/session) and schedule (pre-chemotherapy on day 1 followed by daily sessions on days 2-4) as the true electroacupuncture group.
  Interventions: Device: sham electroacupuncture; Drug: standard quadruple antiemetic therapy

INTERVENTIONS:
Device: electroacupuncture — The acupuncturist applied needles at four acupoints: Zusanli (ST36), Neiguan (PC6), Hegu (LI4), and Zhaohai (KI6), with insertion depths of approximately 20 mm, 15 mm, 20 mm, and 5 mm respectively. Electrical stimulation was delivered in continuous wave mode at 2 Hz frequency with current intensity ≤10 mA (adjusted according to patient tolerance), administered for 30 minutes per session.
  Arms: true acupuncture + standard quadruple antiemetic therapy
Drug: standard quadruple antiemetic therapy — Olanzapine (2.5 mg orally daily, days 1-4), dexamethasone (10 mg intravenously day 1; 7.5 mg intravenously days 2-3), a 5-HT₃ antagonist (palonosetron 0.25 mg intravenously or 0.5 mg orally, or ondansetron 8 mg intravenously or 8 mg orally twice, or tropisetron 5 mg intravenously, all on day 1), and an NK₁ antagonist (fosaprepitant 150 mg intravenously, or aprepitant 130 mg intravenously, or oral aprepitant 125 mg day 1 then 80 mg days 2-3, or netupitant 300 mg orally day 1).
  Arms: true acupuncture + standard quadruple antiemetic therapy
Device: sham electroacupuncture — The same acupoints as the electroacupuncture group were referenced, but with sham acupuncture (minimal insertion at non-acupoint locations) and sham electrical stimulation, while maintaining the same treatment duration and course as the electroacupuncture group.
  Arms: sham acupuncture + standard quadruple antiemetic therapy
Drug: standard quadruple antiemetic therapy — Olanzapine (2.5 mg orally daily, days 1-4), dexamethasone (10 mg intravenously day 1; 7.5 mg intravenously days 2-3), a 5-HT₃ antagonist (palonosetron 0.25 mg intravenously or 0.5 mg orally, or ondansetron 8 mg intravenously or 8 mg orally twice, or tropisetron 5 mg intravenously, all on day 1), and an NK₁ antagonist (fosaprepitant 150 mg intravenously, or aprepitant 130 mg intravenously, or oral aprepitant 125 mg day 1 then 80 mg days 2-3, or netupitant 300 mg orally day 1). All the antiemetic drugs used are the same as those in the true acupuncture group.
  Arms: sham acupuncture + standard quadruple antiemetic therapy

SUMMARY:
This study aims to elucidate the therapeutic efficacy of electroacupuncture in managing chemotherapy-induced gastrointestinal symptom clusters through clinical research. Building upon this foundation, multi-omics analyses will be conducted to investigate the regulatory effects and underlying mechanisms of electroacupuncture on gastrointestinal symptoms. Ultimately, genomic studies will be performed to further clarify the key targets of electroacupuncture intervention, thereby providing high-level evidence-based medical support and theoretical foundations for optimizing electroacupuncture strategies in addressing chemotherapy-induced gastrointestinal symptoms in patients with cancer.

DETAILED DESCRIPTION:
This prospective, multicenter, randomized, double-blind, sham-controlled trial investigates the efficacy of electroacupuncture (EA) combined with standard quadruple antiemetic therapy (olanzapine + dexamethasone + 5-HT3 receptor antagonist + NK-1 receptor antagonist) versus sham EA plus identical antiemetic regimen for chemotherapy-induced gastrointestinal symptom clusters (nausea, vomiting, poor appetite, and xerostomia ). The EA group receives true acupuncture with continuous wave stimulation (2Hz frequency, ≤10mA intensity as tolerated, 30min/session) administered: (1) 1-2h pre-chemotherapy on Day 1, and (2) daily at 9:00-10:00 from Days 2-4. Controls receive sham EA with an identical treatment schedule and the same antiemetics. Assessments during Days 1-5 include: Researchers record the incidence of nausea, vomiting, poor appetite, and xerostomia; Collection of weight, ECOG scores, and EQ-5D-5L questionnaires; documentation of antiemetic/chemotherapy use, concomitant medications, and adverse events; laboratory tests per cycle; and imaging when indicated. Blood samples are preserved every two cycles. Primary/secondary outcomes and adverse events are systematically evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed stage I-III breast cancer;
2. An Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0-1;
3. Age between 18 and 75 years;
4. Scheduled to receive highly emetogenic chemotherapy regimens, such as EC (epirubicin + cyclophosphamide) or platinum-based regimens, during the first cycle of neoadjuvant/adjuvant chemotherapy;
5. No prior acupuncture treatment within one month before enrollment;
6. Voluntary participation in the study with written informed consent obtained; (7) An expected survival of at least 3 months;

(8) Premenopausal women must agree to use contraception during the study period; (9) Adequate bone marrow, liver, and kidney function as defined by standard laboratory criteria.

Exclusion Criteria:

1. Patients with advanced-stage cancer;
2. Those undergoing concurrent chemoradiotherapy;
3. Individuals with severe impairment of vital organ function who cannot tolerate standard-dose chemotherapy;
4. Patients with contraindications to acupuncture, such as active skin infections;
5. Those with digestive system diseases accompanied by nausea and vomiting symptoms that may interfere with accurate assessment;
6. Patients with a history of xerostomia;
7. Individuals with known allergies to the study drugs;
8. Pregnant or breastfeeding patients;
9. Individuals currently using medications with antiemetic activity, such as 5-HT3 receptor antagonists, corticosteroids (except at physiological doses), dopamine receptor antagonists, minor tranquilizers, antihistamines, and benzodiazepines (except for nighttime sedation);
10. Patients with seizure disorders requiring anticonvulsant therapy;
11. Those receiving thiazides as chronic antipsychotic medications;
12. Those with known arrhythmias, uncontrolled congestive heart failure, or acute myocardial infarction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of chemotherapy-induced gastrointestinal symptom clusters, including nausea, vomiting, poor appetite, and xerostomia, within 120 hours after chemotherapy. | 120 hours

SECONDARY OUTCOMES:
Improvement in other gastrointestinal symptom clusters after the first cycle of chemotherapy. | 120 hours
The incidence of no nausea during the acute and delayed phases following the first chemotherapy cycle. | 120 hours
The incidence of no vomiting during the overall, acute, and delayed phases following the first chemotherapy cycle. | 120 hours
Complete response rates in the overall, acute, and delayed phases following the first chemotherapy cycle. | 120 hours
Complete protection rates in the overall, acute, and delayed phases following the first chemotherapy cycle. | 120 hours
Quality of life assessed by the five-level EuroQol five-dimensional questionnaire (EQ-5D-5L). | 120 hours
  The EQ-5D-5L evaluates five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored from 1 ("no problems") to 5 ("extreme problems"), with health states expressed as 5-digit codes (e.g., 11111=no impairment; 55555=extreme impairment across all dimensions). Index scores were calculated using the Chinese value set (Luo et al., 2017), yielding a theoretical range of -0.391 (worse than death) to 1.0 (perfect health). The visual analogue scale (VAS) component records self-rated health status from 0 ("worst imaginable health") to 100 ("best imaginable health").

OTHER OUTCOMES:
Exploratory multi-omics analysis of electroacupuncture's modulation on symptom clusters. | From enrollment through the entire chemotherapy cycle (up to 8 cycles, each cycle is 21 days; maximum 64 weeks)
Association between electroacupuncture and pathological complete response rate in patients receiving neoadjuvant therapy. | From enrollment through the entire chemotherapy cycle From enrollment through the entire chemotherapy cycle (up to 8 cycles, each cycle is 21 days; maximum 64 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Qinghai University Affiliated Hospital, Xining, Qinghai, China